CLINICAL TRIAL: NCT07211594
Title: HEALTH-RELATED QUALITY OF LIFE OF ADOLESCENTS WITH CEREBRAL PALSY: AGREEMENT BETWEEN ADOLESCENTS, CAREGIVERS AND PHYSIOTHERAPISTS
Brief Title: HEALTH-RELATED QUALITY OF LIFE IN CEREBRAL PALSY: AGREEMENT BETWEEN ADOLESCENTS, CAREGIVERS AND PHYSIOTHERAPISTS
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Mintaze Kerem Gunel, Prof. Dr., Hacettepe University
Other Study IDs: GO 18/876-02
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Health-Related Quality-of-Life; Adolescent; Cerebral Palsy (CP)
Keywords: health-related quality of life; cerebral palsy (CP); adolescent
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adolescents with cerebral palsy: The study was conducted with 97 adolescents CP attending Hacettepe University Physiotherapy and Rehabilitation Department's Pediatric Rehabilitation together with their caregivers.
- Caregivers of adolescent with cerebral palsy: Caregivers of adolescent with cerebral palsy who may be parents, grandparents or caregivers.
- the physiotherapist who conducts the adolescent rehabilitation process.: pediatric physiotherapists working in the field of pediatric rehabilitation especially with cerebral palsy

SUMMARY:
Health-related quality of life (HRQoL) has recently become a widely used outcome measure. Although self-reporting is considered the gold standard, proxy reports are commonly used for adolescents with cerebral palsy (CP).

Study Question: Is there agreement between adolescents, caregivers and physiotherapists in health-related quality of life reports in adolescents with cerebral palsy?

DETAILED DESCRIPTION:
Cerebral palsy are often accompanied by sensory, perceptual, developmental, and behavioral problems, as well as epilepsy and secondary musculoskeletal disorders. As a result of these impairments, children and adolescents with CP have functional limitation that affect their daily lives. These limitations adversely affect their quality of life depending on the severity of functional impairments. Health-related quality of life is conceptualized as an individual's subjective evaluation of life domains that are perceived to be influenced by a medical condition or its treatment. Informed by the International Classification of Functioning, Disability and Health (ICF) and the socio-ecological model, the primary aim of interventions for individuals with cerebral palsy and their families should be to enhance quality of life. Previous research has shown that the level of agreement on HRQoL between physicians and adolescents is generally lower than that between parents and adolescents. When the caregiver is more familiar with the adolescent with CP-such as a parent rather than a medical professional-the likelihood of agreement between the adolescent and the caregiver tends to be higher. Agreement on target problems is essential for effective treatment planning. Differences between adolescents and their caregivers can influence treatment decisions; thus, combining self- and proxy-reports offers a more comprehensive assessment of HRQoL. Therefore, a multi-informant approach, considered the gold standard in CP research and practice, integrates reports from children, parents, and when appropriate professionals such as teachers or clinicians, providing a comprehensive assessment of the child's quality of life across different contexts.

Another important issue in measuring quality of life in individuals with CP is that the scales used should address CP-specific concerns. Therefore, using CP-specific measurement tools is recommended to provide clearer outcomes for intervention processes. Although research has compared the quality of life perspectives of children and adolescents with CP and their parents, there remains a lack of studies investigating the agreement between reports from adolescents with CP, their parents, and the professionals involved in their care. The main objective of this study is to assess the agreement and differences between the views of adolescents with CP, their families.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with CP of all clinical types,
* aged 11-18 years,
* who can understand and answer the questions.

Exclusion Criteria:

* Adolescents who did not attend regular therapy sessions
* Physiotherapists who performed therapy sessions with the adolescent for less than four weeks

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The demographic information such as weight, height, sex, age etc. were recorded for adolescents, as well as the age and educational status of the caregivers. Gross Motor Function Classification System (GMFCS-E&R) were used to classify the adolescents' gross motor function. The hand function of adolescents in daily activities was classified with The Manual Ability Classification System (MACS), and the communication of adolescents was classified with the Communication Function Classification System (CFCS). Clinicians and researchers used these classification systems to grade functional capacity systems and constitute a common language to describe function.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2019-05-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Health-Related Quality of Life: The Pediatric Quality of Life Inventory (PedsQL) Measurement Tool | 5-10 minutes
  PedsQL was designed to evaluate HR-QOL in generic and disease-specific situations with disease-specific modules in children and adolescents between 2-18 years old. The PedsQL 3.0 CP Module was designed to measure HR-QOL dimensions specific to CP. PedsQL 3.0 CP encompasses 35-item in Module seven scales: (1) Daily Activities (9 items); (2) School Activities (4 items); (3) Movement and Balance (5 items); (4) Pain and Hurt (4 items); (5) Fatigue (4 items); (6) Eating Activities (5 items); and (7) Speech and Communication (4 items). The Scales are included in parallel adolescent self-report and parent proxy-report formats. A 5-point Likert scale is used across adolescent self-reports for ages 8 to 18 years and parent proxy reports (0=never a problem; 1=almost never a problem; 2=sometimes a problem; 3=often a problem; 4=almost always a problem). Items are reverse scored and transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0) so that higher scores indicate better HRQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Mintaze Kerem Gunel, Prof. Dr., Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Sentenac M, Rapp M, Ehlinger V, Colver A, Thyen U, Arnaud C. Disparity of child/parent-reported quality of life in cerebral palsy persists into adolescence. Dev Med Child Neurol. 2021 Jan;63(1):68-74. doi: 10.1111/dmcn.14638. Epub 2020 Jul 25. PMID 32710687
- [Background] Morrow AM, Hayen A, Quine S, Scheinberg A, Craig JC. A comparison of doctors', parents' and children's reports of health states and health-related quality of life in children with chronic conditions. Child Care Health Dev. 2012 Mar;38(2):186-95. doi: 10.1111/j.1365-2214.2011.01240.x. Epub 2011 Jun 8. PMID 21651605
- [Background] Aza A, Riquelme I, Gomez Vela M, Badia M. Proxy- and self-report evaluation of quality of life in cerebral palsy: Using Spanish version of CPQOL for Children and adolescents. Res Dev Disabil. 2024 Nov;154:104844. doi: 10.1016/j.ridd.2024.104844. Epub 2024 Sep 24. PMID 39321691